CLINICAL TRIAL: NCT01924663
Title: Viral Illness in the Pediatric Critical Care Setting: the Incidence, Timing and Severity of Associated Myocardial Dysfunction and Acute Kidney Injury.
Brief Title: Viral Illness in Pediatric Critical Care: Incidence Timing & Severity of Associated Heart Dysfunction & Acute Kidney Injury
Acronym: MyDAKI-01
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Tanya Holt, Principal Investigator, Director of Paediatric Critical Care, University of Saskatchewan
Other Study IDs: MyDAKI-01
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure; Acute Kidney Injury
Keywords: Heart Failure; Acute Kidney Injury; Myocardial Dysfunction; Pediatric Critical Care; Pediatric Intensive Care Units; Respiratory Virus
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to be able to better describe the incidence, timing and severity of myocardial dysfunction and acute kidney injury (AKI) following a documented respiratory viral illness (RSV, adenovirus, metapneumovirus, parainfluenza, influenza, etc.) in pediatric patients.

DETAILED DESCRIPTION:
This is a single-centre, prospective and retrospective, descriptive data-collection pilot study.

Prospective Data Collection:

All pediatric patients who are less than 18 years with a confirmed positive respiratory viral swab will be invited to participate.

Retrospective Data Collection:

The retrospective portion of this study will examine a 5 year period prior to the start of enrollment for the prospective study, with the intention to include all pediatric patients who are less than 18 years with a confirmed positive respiratory viral swab and admitted into the local hospital's PICU.

ELIGIBILITY:
Inclusion Criteria:

1. The parent or legal guardian of the pediatric subject must sign the Consent Form for participants in the prospective portion of the study.
2. The subject must be no greater than 18 years of age, at the time of consent.
3. The subject must be admitted to the local hospital.
4. The subject must have a confirmed positive respiratory viral swab.

Exclusion Criteria:

1. The parent or legal guardian of the pediatric subject is unavailable or unwilling to sign the Consent Form for participants in the prospective portion of the study.
2. The subject has had previous kidney injury or myocardial dysfunction prior to positive respiratory viral swab.
3. The subject has any previous problems (prior to positive respiratory viral swab) with their heart or kidneys that could compromise the results, in the opinion of the Investigator.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric subjects admitted to the local hospital with a confirmed positive respiratory viral swab.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Myocardial dysfunction, as defined by a low ejection fraction on an Echocardiogram. | up to 7 days
Acute Kidney Injury (AKI) as defined by the meeting of the pediatric RIFLE criteria. | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Holt, M.D., Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada